CLINICAL TRIAL: NCT03121755
Title: CCK1R Function in Patient Leukocytes
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Laurence J. Miller, Professor of Biochemistry and Molecular Biology and Medicine and Pharmacology, Mayo Clinic
Other Study IDs: 15-000131
Record Dates: First submitted 2017-04-17; First posted 2017-04-20 (Actual); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Obesity; Diabetes Mellitus, Type 2; Metabolic Syndrome
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sangre Por Salud cohort members: Subjects entered in the Sangre Por Salud Biobank

SUMMARY:
The type 1 cholecystokinin receptor (CCK1R) is a potential target for the treatment of obesity, due to the ability of this GI hormone to elicit satiety. However, this receptor has been shown to be sensitive to the cholesterol content of the membrane in which it is expressed. Because some patients who might be candidates for the use of CCK agonists to treat their obesity and co-morbidities, the goal of this study is to determine how metabolic abnormalities might affect the responsiveness of this receptor to CCK. Because the normal site mediating CCK-stimulated satiety is on vagal afferent neurons that cannot easily be studied, we will collect buffy coat cells from a peripheral blood sample from patients involved in the Sangre Por Salud Biobank at Mountain Park Medical Center. Ex vivo, the CCK1R will be expressed on these cells and will be functionally characterized, and the cholesterol content of the cells will be assayed. These data will be correlated with the clinical, biochemical, and metabolic phenotypic data collected as part of the parent study.

DETAILED DESCRIPTION:
Subjects are volunteers who provide prospective informed consent to be entered into the Sangre Por Salud Biobank at Mountain Park Medical Center. These include men and women age 18-85 of Hispanic/Latino descent, who are not pregnant or have given birth in the previous 12 months, or who are nursing, and who have not been diagnosed with cancer in the previous three years. Two groups of patients are included, representing those who have not been diagnosed as having diabetes, and those with diabetes. Subjects undergo entry physical examination and standard metabolic phenotyping, with the non-diabetics also undergoing a 2-hour glucose tolerance test. Blood samples are also banked and available for other studies, such as the one now being described.

For the current study, 5 ml of blood will be coded and delivered in an anonymized form. Buffy coat cells will be isolated and infected ex vivo with a viral construct including the wild type CCK1R tagged with a fluorescent tag. Cells will be placed in culture overnight and harvested for quantitation of receptor expression and determination of CCK responsiveness and cholesterol content. These data will be correlated with selected relevant clinical, biochemical, and morphometric data.

ELIGIBILITY:
Inclusion Criteria:

* volunteers

Exclusion Criteria:

* Hispanic/Latino descent not pregnant, or given birth in the previous 12 months, or currently nursing not diagnosed with cancer in the past three years

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: subjects in Sangre Por Salud Biobank
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2015-01-21 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-04-14 (Actual)

PRIMARY OUTCOMES:
Total cellular cholesterol on leukocytes collected from the subjects | baseline
  The cells will be lysed by sonication; neutral sterols will be extracted, and the cholesterol will be quantified using an assay.

CONTACTS AND LOCATIONS:
Overall Officials: Laurence J Miller, MD, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Desai AJ, Dong M, Langlais BT, Dueck AC, Miller LJ. Cholecystokinin responsiveness varies across the population dependent on metabolic phenotype. Am J Clin Nutr. 2017 Aug;106(2):447-456. doi: 10.3945/ajcn.117.156943. Epub 2017 Jun 7. PMID 28592602